CLINICAL TRIAL: NCT04297618
Title: The Effect of Xiidra on Comfort and Dryness in Symptomatic Contact Lens Wearers
Acronym: COLLIE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 41189
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2024-06

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — lifitegrast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Xiidra treatment (Experimental): Each participant will use the same study drops, Xiidra, over the course of the 12-week study.
  Interventions: Drug: Xiidra

INTERVENTIONS:
Drug: Xiidra — Xiidra (lifitegrast 5% ophthalmic solution)
  Other Names: Lifitegrast

SUMMARY:
The purpose of this study to evaluate changes in comfort and dryness in symptomatic contact lens (CL) wearers after using Xiidra (lifitegrast 5.0% ophthalmic solution) for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 18 years of age and has full legal capacity to volunteer;
2. Has read and signed an information consent letter;
3. Is willing and able to follow instructions and maintain the appointment schedule;
4. Currently wears daily, soft, frequent replacement lenses (daily, bi-weekly or monthly disposable lenses) in both eyes, that are available in Canada, for a minimum of 5 days/week for 6 hours/day over the last month, and is willing to continue to do so during the study;
5. Is a symptomatic CL wearer as determined by Eye Dryness Score4,5 (EDS) ≥40 at the end of the wear day AND according to the classification by Young et al7;
6. Can achieve acceptable lens fit as well as visual acuity (VA) correctable to logMAR +0.20 or better in each eye with their habitual contact lens type;
7. Has a history of artificial tear or rewetting drop use at least once in the last 30 days;
8. Is willing to use the Xiidra study drops twice a day on a daily basis (irrespective of CL wear) and to stop use of any habitual rewetting drops and/or artificial tears over the course of the 12-week treatment phase;

Exclusion Criteria:

1. Is participating in any concurrent clinical or research study;
2. Is wearing soft CLs on an extended wear basis (i.e. overnight) or is a rigid gas permeable lens or hybrid lens wearer;
3. Has a known sensitivity to the investigational product or diagnostic substances (e.g. fluorescein) to be used in the study;
4. Has any known ocular disease and/or infection, that's either currently active* or has occurred within the previous 30 days;
5. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable (examples may include active or uncontrolled systemic conditions such as allergies, autoimmune disease or immunodeficiency disease);
6. Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable, including but not limited to topical cyclosporine, any other topical ophthalmic medication, antihistamines, and aspirin;
7. Is pregnant, lactating or planning a pregnancy at the time of enrolment (by self-report);**
8. Has undergone refractive error surgery such as LASIK within the last 12 months;
9. Has a history of yttrium-aluminium-garnet laser posterior capsulotomy within the previous 6 months,
10. Is an employee of the Centre for Ocular Research & Education; * For the purposes of this study, active ocular disease is defined as infection or inflammation which requires therapeutic treatment. Mild (i.e. not considered clinically relevant) lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining and dry eye are not considered active ocular disease. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD, FCOptom, Principal Investigator — Centre for Ocular Research & Education
Locations (1):
- Centre for Ocular Research & Education, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at a single site between July 2021 and April 2024. The first participant was enrolled on July 7, 2021 and the last participant was enrolled January 19, 2024.
Pre-assignment Details: Out of the 45 participants that were enrolled, 43 met the inclusion critieria, and 42 were dispensed with the study treatment.
Period: Overall Study
Arm/Group | Xiidra Treatment
Started | 42
Completed | 40
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All suitable participants who were eligible to take part in the study.
Arm/Group | Xiidra Treatment
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 43

OUTCOME MEASURES:

1. Primary Outcome: Difference in Contact Lens-related Discomfort at 12 Weeks Compared to Baseline
Description: Participants rate their contact lens-related discomfort on a scale from 0 (no discomfort) to 100 (maximal discomfort).
Time Frame: Baseline and 12 weeks
Population: 2 participants discontinued before the study could be completed.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Xiidra Treatment
Number analyzed (Participants) | 40
score on a scale
  Baseline | 71 [8 to 93]
  12 Weeks | 11 [0 to 96]
Statistical Analysis 1: Comparison: Xiidra Treatment; Test type: Other; p < 0.01, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Difference in Contact Lens-related Dryness at 12 Weeks Compared to Baseline
Description: Participants rate their contact lens-related dryness on a scale from 0 (no discomfort) to 100 (maximal discomfort).
Time Frame: Baseline and 12 weeks
Population: 2 participants discontinued before the study could be completed.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Xiidra Treatment
Number analyzed (Participants) | 40
score on a scale
  Baseline | 75 [40 to 96]
  12 Weeks | 15 [0 to 98]
Statistical Analysis 1: Comparison: Xiidra Treatment; Test type: Other; p < 0.01, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Regular investigator assessment
Groups:
- Ocular Adverse Events (After Xiidra Was Dispensed): Ocular adverse events in all participants who were dispensed with the study product.
- Systemic Adverse Events (After Xiidra Was Dispensed): Systemic adverse events in all participants who were dispensed with the study product.
- Ocular Adverse Events (Before Xiidra Was Dispensed): Ocular adverse events that occurred in all participants that were eligible for the study prior to the study product being dispensed.
- Systemic Adverse Events (Before Xiidra Was Dispensed): Systemic adverse events that occurred in all participants that were eligible for the study prior to the study product being dispensed.
Arm/Group | Ocular Adverse Events (After Xiidra Was Dispensed) | Systemic Adverse Events (After Xiidra Was Dispensed) | Ocular Adverse Events (Before Xiidra Was Dispensed) | Systemic Adverse Events (Before Xiidra Was Dispensed)
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42 | 1/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42 | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 3/42 | 6/42 | 1/43 | 0/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocular Adverse Events (After Xiidra Was Dispensed) (N=42) | Systemic Adverse Events (After Xiidra Was Dispensed) (N=42) | Ocular Adverse Events (Before Xiidra Was Dispensed) (N=43) | Systemic Adverse Events (Before Xiidra Was Dispensed) (N=43)
Irritated, red eye & purulent discharge (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial conjunctivitis (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Bacterial conjunctivitis/Acute bacterial conjunctivitis
Watery eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Teary (watery) eye
COVID (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — COVID
Leukocytoclastic vasculitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dryness around periorbital eyelid skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corneal sterile infiltrates (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Infiltrative keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/18/NCT04297618/Prot_SAP_000.pdf